CLINICAL TRIAL: NCT06763029
Title: Phase II Exploratory Study of Irinotecan Liposomes Combined with Cetuximab + Vermofenib in First-line Failure of Advanced RAS Wild /BRAF Mutated Colorectal Cancer
Brief Title: Irinotecan Liposomes Combined with Cetuximab + Vermofenib in First-line Failure of Advanced Colorectal Cancer
Acronym: VICPROIRI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Li Wenhua, Internal Medicine oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FudanU.2411307-18
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal cancer; Irinotecan liposomes; BRAF V600E mutation; Vermofenib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Intervention Model Description: Single-center, single-arm, prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Irinotecan liposome gourp (Experimental): Irinotecan liposomes combined with cetuximab + vermofenib
  Interventions: Drug: Irinotecan liposomes combined with cetuximab + vermofenib

INTERVENTIONS:
Drug: Irinotecan liposomes combined with cetuximab + vermofenib — Vermofenil 960mg orally twice daily; Irinotecan liposomes, 70mg/m2, d1, 90 min intravenously, Q2W; Cetuximab 500mg/m2, d1, Q2W;
  Other Names: Irinotecan liposomes+VC

SUMMARY:
Efficacy and safety of irinotecan liposomes combined with cetuximab + vermofenib in first-line failure of advanced RAS wild /BRAF mutated colorectal cancer, Exploratory analysis of biomarkers (including but not limited to ctDNA, immune microenvironment indicators, tumor mutation load, lymphocyte subsets, cytokines, gut microbes, and others) in relation to efficacy.

DETAILED DESCRIPTION:
This study aims to explore the following key questions: 1) whether replacing ordinary irinotecan in VIC protocol with irinotecan liposomes can improve the safety and efficacy of BRAF V600E mutation in second-line treatment of metastatic colorectal cancer; 2) To provide a reference for identifying the dominant population for the benefit of irinotecan liposomes through the exploration of a range of biomarkers (including but not limited to ctDNA, immune microenvironmental indicators, tumor mutation load, lymphocyte subsets, cytokines, gut microbes, and others). Thus, it provides more treatment options for BRAF V600E mutations in patients with metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age;
* Colorectal adenocarcinoma was confirmed by histological or cytopathological examination, and RAS wild /BRAF V600E mutation was detected by PCR or NGS;
* Failure or intolerance of standard first-line treatment. First-line regimens including oxaliplatin and/or irinotecan in combination with fluorouracil in patients with MSS; For BRAF V600E mutated patients with MSI-H, first-line immunotherapy with PD-1 or PD-L1 is required;
* At least one measurable lesion according to RECIST v1.1;
* ECOG score is 0~2;
* Good bone marrow and organ function: ① Neutrophils (ANC) ≥1.5×109/L, platelets (PLT) ≥100×109/L, hemoglobin (Hb) ≥90g/L, white blood cells (WBC) ≥3.0×109/L, albumin (ALB) ≥32 g/L, and no bleeding tendency; ② AST, ALT and alkaline phosphatase (ALP) were all ≤2.5× upper limit of normal range (ULN), and ≤5×ULN when liver metastases occurred; Total bilirubin ≤1.5×ULN; Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60 ml/min (calculated according to Cockroft-Gault);
* Expected survival ≥3 months;
* Can understand the situation of this study, patients and (or) legal representatives voluntarily agree to participate in this study and sign informed consent.

Exclusion Criteria:

* Patients who have previously received BRAF inhibitors or irinotecan liposomes;
* Proven allergic to the test drug and/or its excipients;
* symptomatic, untreated brain metastases or meningeal metastases that fail to achieve clinical stability;
* Acute or subacute intestinal obstruction or chronic inflammatory bowel disease;
* have had other malignant tumors within the past 5 years or currently, except for cured cervical carcinoma in situ, uterine carcinoma in situ and non-melanoma skin cancer;
* Pregnant or lactating female patients, patients of childbearing age who refuse to accept contraceptive measures;
* Patients considered by the investigator to be unsuitable for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | The evaluation period was up to 24 months from the date the participant entered the clinical study and started the medication
  The proportion of patients with optimal tumor response, complete response (CR) or partial response (PR) assessed based on the RECIST v1.1 criteria

SECONDARY OUTCOMES:
Progression free survival | The evaluation period was up to 24 months from the date of the subject's first medication to the date of first recorded progress or the date of death from any cause, whichever came first
  The time from the start of treatment to the first recording of PD or death, whichever occurs first
Overall survival | The evaluation period was up to 24 months from the date of the subject's first medication to the date of death from any cause
  The time between the start of treatment and the first recorded death
Adverse event | Incidence and severity of adverse events in treatment regimens up to 24 months
  Incidence and severity of adverse events in treatment regimens

CONTACTS AND LOCATIONS:
Overall Officials: Wenhua Li, Ph.D, Principal Investigator — Affiliated Cancer Hospital of Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
After the research is completed, it is decided to share according to the research results